CLINICAL TRIAL: NCT04073329
Title: Assessing Postoperative Reduction Following Acetabular Fracture Surgery
Brief Title: Acetabular Fracture Reduction Assessment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bahaaeldin Mohamed Abdelhafez, Principal investigator, Assiut University
Other Study IDs: AFRA
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Acetabular Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Plain x ray: measurement the accuracy of post operative reduction by Matta method
  Interventions: Other: post operative measure of reduction
- CT: measure the accuracy of reduction by Verbeek method
  Interventions: Other: post operative measure of reduction

INTERVENTIONS:
Other: post operative measure of reduction — measurement was used to grade quality of reduction according to Matta's system . In accordance with prior studies, adequate (or anatomic) reductions with 0-1 mm of displacement were compared to inadequate (imperfect or poor) reductions with > 1 mm displacement . For the CT-based method, postoperative pre-digital (prior to 2000) and digital CT images were independently assessed in the axial, sagittal, and coronal planes, and residual gap and step displacement were measured along the articular surface at the level of the weight-bearing dome. Adequate reductions on postoperative CT were defined as < 1 mm step and < 5 mm gap displacement and inadequate reductions as ≥ 1 mm step and/or ≥ 5 mm gap displacement.

SUMMARY:
It is widely accepted in the literature that quality of acetabular fracture reduction is one of the most important factor for the outcome. To obtain best results, anatomical reduction has to be obtained. Intra-operative radiographic assessment depends mainly on plain x-ray. Plain x-ray alone is not enough for post-operative assessment as it depends mainly on reduction of the dome with concentricity of the hip.

DETAILED DESCRIPTION:
It is widely accepted in the literature that quality of acetabular fracture reduction is one of the most important factor for the outcome. To obtain best results, anatomical reduction has to be obtained. Intra-operative radiographic assessment depends mainly on plain x-ray. Plain x-ray alone is not enough for post-operative assessment as it depends mainly on reduction of the dome with concentricity of the hip. Complex fractures with multi-fragmentary fracture pattern, impacted fragments (marginal or roof), fractures with osteo-chondral loss and associated head of femur injuries, pose problems with reduction assessment using both Plain x-ray and CT due to lack of clear standardized way of assessment. Matta criteria has been used widely in the literature for assessment, however it lacks some important criteria which directly related to the functional outcome. Few papers in the literature address this problem and reporting some ways for assessment but with lack of testing and reproducibility.

Since there is in our level 1 trauma center a lot of cases of acetabular fractures that is admitted yearly to our center Purpose of our study is to use those methods for our cases in order to test their validity and reproducibility

ELIGIBILITY:
Inclusion Criteria:

* Isolated displaced acetabular fractures
* Skeletally mature patients

Exclusion Criteria:

* Skeletally Immature

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients included in our study will have postoperative plain X-rays and comparing it to CT scan to assess their quality of reduction and other criteria mentioned in the literature.
  10 observers with different years of experience will assess all fractures using plain x-ray and CT.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Ability of CT scans and plain radiographs to detect residual articular steps and gaps after healing of acetabular fractures managed by open reduction and internal fixation. | 1 year
  measurement was used to grade quality of reduction according to Matta's system . In accordance with prior studies, adequate (or anatomic) reductions with 0-1 mm of displacement were compared to inadequate (imperfect or poor) reductions with > 1 mm displacement . For the CT-based method, postoperative pre-digital (prior to 2000) and digital CT images were independently assessed in the axial, sagittal, and coronal planes, and residual gap and step displacement were measured along the articular surface at the level of the weight-bearing dome. Adequate reductions on postoperative CT were defined as < 1 mm step and < 5 mm gap displacement and inadequate reductions as ≥ 1 mm step and/or ≥ 5 mm gap displacement.

REFERENCES:
- [Background] Borrelli J Jr, Ricci WM, Steger-May K, Totty WG, Goldfarb C. Postoperative radiographic assessment of acetabular fractures: a comparison of plain radiographs and CT scans. J Orthop Trauma. 2005 May-Jun;19(5):299-304. PMID 15891537
- [Background] Verbeek DO, van der List JP, Helfet DL. Computed tomography versus plain radiography assessment of acetabular fracture reduction is more predictive for native hip survivorship. Arch Orthop Trauma Surg. 2019 Dec;139(12):1667-1672. doi: 10.1007/s00402-019-03192-w. Epub 2019 Apr 27. PMID 31030241
- [Background] Dodd A, Osterhoff G, Guy P, Lefaivre KA. Radiographic Measurement of Displacement in Acetabular Fractures: A Systematic Review of the Literature. J Orthop Trauma. 2016 Jun;30(6):285-93. doi: 10.1097/BOT.0000000000000538. PMID 27206254